CLINICAL TRIAL: NCT06571383
Title: Weight Maintenance in Adolescents With Obesity; Long-Term Treatment With Semaglutide s.c.2.4 mg Once-weekly
Brief Title: STEP TEENS Weight Maintenance: A Research Study on How Well Semaglutide Helps Teenagers With Excess Body Weight to Lose Weight and Maintain Weight Loss
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN9536-7752; U1111-1295-4799 (Other: World Health Organisation (WHO)); 2023-508055-40 (Other: European Medical Agency (EMA))
Record Dates: First submitted 2024-08-22; First posted 2024-08-26 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Semaglutide (Experimental): 2.4mg or maximum tolerated dose(MTD) injected subcutaneously (under the skin, s.c) once weekly
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: Semaglutide — Participants will receive semaglutide s.c(under the skin) once weekly.

SUMMARY:
The study is testing how well semaglutide can help adolescents with excess body weight to lose weight and to maintain weight loss. All participants in the study will receive semaglutide as a weekly injection. The study medicine is injected with a thin needle in the stomach, thighs or upper arms. All participants will get semaglutide treatment for a minimum of 3 years.

ELIGIBILITY:
Inclusion criteria:

* Informed consent obtained before any study-related activities. Study-related activities are any procedures that are carried out as part of the study, including activities to determine suitability for the study:

  1. The parent(s) or legally acceptable representative (LAR) of the participant must sign and date the Informed Consent Form, according to local requirements
  2. The participant must sign and date the Child Assent Form or provide oral assent, according to local requirements
* Age 12 to less than 15 years at the time of signing the informed consent
* BMI greater than or equal to 95th percentile at screening
* Body weight greater than 60 kg at screening

Exclusion criteria:

* Prepubertal status (Tanner stage 1)
* Treatment with any medication prescribed for the indication of obesity or weight management within 90 days before screening
* Previous or planned (during the study period) obesity treatment with surgery or a weight loss device. However, the following are allowed:

  1. Liposuction and/or abdominoplasty, if performed more than 1 year prior to screening
  2. Adjustable gastric banding, if the band has been removed more than 1 year prior to screening
  3. Intragastric balloon, if the balloon has been removed more than 1 year prior to screening
  4. Duodenal-jejunal bypass liner (e.g., Endobarrier), if the sleeve has been removed more than 1 year prior to screening
* Endocrine, hypothalamic, or syndromic obesity
* History of type 1 or type 2 diabetes mellitus

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 500 (Estimated)
Dates: Start 2024-09-17 (Actual); Primary Completion 2028-11-15 (Estimated); Study Completion 2031-11-15 (Estimated)

PRIMARY OUTCOMES:
Maintenance of Body Mass Index (BMI) below obesity threshold | From 1.5 years to 3 years
  Measures as count of participants

SECONDARY OUTCOMES:
Maintenance of improved Body Mass Index (BMI) category | From 1.5 years to 3 years and end of continued treatment phase (up to 6 years)
  Measured as count of participants
Tapering to zero dose | From 1.5 years to 3 years
  Measured as count of participants
Time/dose steps before ending dose tapering | From 1.5 years to 3 years
  Measured in weeks, count of dose steps
Achieving Body Mass Index (BMI) below obesity threshold | From baseline (day 0) to 1.5, 3 years and end of continued treatment phase (up to 6 years)
  Measured as count of participants
Achieving any improvement in Body Mass Index (BMI) category | From baseline (day 0) to 1.5, 3 years, and end of continued treatment phase (up to 6 years)
  Measured as count of participants
Change in Body Mass Index (BMI) | From baseline (day 0) to 1.5 and 3 years
  Measured in percentage (%)
Body Mass Index (BMI) percentage of the 95th percentile | From baseline (day 0) to 1.5 and 3 years
  Measured in percentage (%)
Change in Body Mass Index Standard Deviation Score (BMI SDS) | From baseline (day 0) to 1.5 and 3 years
  Unitless
Change in waist-to-height ratio (waist [cm]/ height [cm]) | From baseline (day 0) to 1.5 and 3 years
  Unitless
Change in waist circumference | From baseline (day 0) to 1.5 and 3 years
  Measured in centimeters (cm)
Change in HbA1c | From baseline (day 0) to 1.5, 3 years and end of continued treatment phase (up to 6 years)
  Measured in percentage (%) points
Change in fasting plasma glucose | From baseline (day 0) to 1.5, 3 years and end of continued treatment phase (up to 6 years)
  Measured in millimol per liter (mmol/L), milligram per deciliter (mg/dL)
Change in fasting insulin and Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) | From baseline (day 0) to 1.5, 3 years and end of continued treatment phase (up to 6 years)
  Measured in percentage (%)
Change in high sensitivity C-reactive protein (hsCRP) | From baseline (day 0) to 1.5, 3 years and end of continued treatment phase (up to 6 years)
  Measured in percentage (%)
Change in alanine aminotransferase (ALT), total cholesterol, high density lipoprotein (HDL), low density lipoprotein (LDL), very low-density lipoprotein (VLDL) and triglycerides | From baseline (day 0) to 1.5, 3 years and end of continued treatment phase (up to 6 years)
  Measured in percentage (%)
Change in systolic and diastolic blood pressure | From baseline (day 0) to 1.5, 3 years and end of continued treatment phase (up to 6 years)
  Measured in millimetres of mercury (mmHg)
Change in fat mass, by dual X-ray absorptiometry (DXA) relative to total body mass | From baseline (day 0) to 1.5 and 3 years
  Measured in percentage (%) points
Change in lean body mass, by dual X-ray absorptiometry (DXA) relative to total body mass | From baseline (day 0) to 1.5 and 3 years
  Measured in percentage (%) points
Relative change in visceral fat mass, by dual X-ray absorptiometry (DXA) | From baseline (day 0) to 1.5 and 3 years
  Measured in percentage (%)
Serious Adverse Event (SAE) | From baseline (day 0) to 1.5 years, from 1.5 to 3 years, and from 3 years to end of continued treatment phase (up to 6 years)
  Count

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (93):
- United States (26):
  - Neighborhood Healthcare, Escondido, California
  - Clinical Neuroscience Solution, Orlando, Florida
  - TMH Physician Partners Endo, Tallahassee, Florida
  - Children's Healthcare Atlanta, Atlanta, Georgia
  - Columbus Research Foundation, Columbus, Georgia
  - Eastside Bariatric and Gen Surg, Snellville, Georgia
  - Solaris Clinical Research, Meridian, Idaho
  - Synexus Clinical Research US Inc.-Chicago, Chicago, Illinois
  - Indiana University Hospital, Indianapolis, Indiana
  - University Of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Pennington Biom Res Ctr, Baton Rouge, Louisiana
  - Barry J. Reiner, MD LLC, Baltimore, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - Mississippi CTR for ADV MED, Madison, Mississippi
  - UBMD Peds-Div of Endo/Diabetes, Buffalo, New York
  - WakeMed Childn Endo-Dbt_Raleig, Raleigh, North Carolina
  - Valley Weight Loss Clinic, Fargo, North Dakota
  - Centricity Research - Ohio, Columbus, Ohio
  - PriMed Clinical Research, Dayton, Ohio
  - UPMC Child Hosp-Pittsburgh, Pittsburgh, Pennsylvania
  - Coastal Carolina Research Ctr, North Charleston, South Carolina
  - Clinical Neuroscience Solutions, Memphis, Tennessee
  - Texas Diabetes Institute, San Antonio, Texas
  - Clinical Trials of Texas Inc, San Antonio, Texas
  - Health Res of Hampton Roads, Newport News, Virginia
  - Virginia Commonwealth Univ, Richmond, Virginia
- Belgium (4):
  - UZ Brussel - Universitair Ziekenhuis Brussel, Brussels
  - Cliniques universitaires Saint-Luc, Brussels
  - UZA - Universitair Ziekenhuis Antwerpen, Edegem
  - Uz Leuven, Leuven
- Canada (8):
  - Alberta Children's Hospital, Calgary, Alberta
  - Stollery Children's Hospital, Edmonton, Alberta
  - BC Children's Hospital, Vancouver, British Columbia
  - Markham Stouffville Hosp, Markham, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - McMaster Children's Hospital, West Hamilton, Ontario
  - Maison de Sante Prevention, Montreal, Quebec
  - McGill Uni Health Ctre - Glen Site, Montreal, Quebec
- Denmark (3):
  - Aalborg Universitetshospital, Aalborg
  - Aarhus Universitetshospital, Steno Diabetes Center Aarhus, Aarhus
  - Holbæk Sygehus - Børne- og Ungeafdelingen, Holbæk
- France (5):
  - Centre Hospitalier Universitaire de Lille-Hopital Jeanne de Flandre, Lille
  - Fondation Lenval Nice, Nice
  - Ap-Hp_Hopital Armand Trousseau, Paris
  - Centre Hospitalier Universitaire de Rouen-Hopital Charles Nicolle, Rouen
  - Hopital Des Enfants, Toulouse
- Germany (9):
  - Kath. Klinikum Bochum gGmbH - Kinderklinik St. Josef-Hospital, Bochum
  - Uni-Med. Göttingen - Klinik für Kinder- und Jugendmedizin, Göttingen
  - Universitätsmedizin Göttingen - Klinik für Kinder-und Jugendmedizin, Göttingen
  - Auf der Bult - Klinik für Diabetologie, Endokrinologie, Gastroenterologie und Klinische Forschung, Hanover
  - Hannoversche Kinderheilanstalt "Auf der Bult" - Diabeto-, Endokrino-, Gastroenterologie und Klinische Forschung, Hanover
  - Uniklinik Leipzig - Klinik und Poliklinik für Kinder- und Jugendmedizin, Leipzig
  - Universitätsklinikum Leipzig - Klinik und Poliklinik für Kinder- und Jugendmedizin, Leipzig
  - Uniklinik Ulm - Dt. Zentrum für Kinder- und Jugendgesundheit (DZKJ), Ulm
  - Universitätsklinikum Ulm für Kinder- und Jugendmedizin, Ulm
- Greece (5):
  - U.G.H. "Attikon", Pediatric Endocrinology Outpatient Clinic, Athens
  - P & A Kyriakou Childrens' Hospital, Goudi/Athens
  - General University of Patra - Paediatric Department, Pátrai
  - 'Ippokrateio' General Hospital of Thessaloniki, Thessaloniki
  - Ippokrateio Gen Hosp of Thessaloniki, 1st Pediatric Clinic, Thessaloniki
- Italy (5):
  - IRCCS Meyer Firenze, Florence, Tuscany
  - Ospedale dei Bambini "Vittore Buzzi", Milan
  - Ospedale Pediatrico Bambino Gesu, Roma
  - IRCCS materno infantile Burlo Garofolo - Clinica Pediatrica, Trieste
  - Azienda Ospedaliera Universitaria Integrata Verona - Ospedale Civile Maggiore Borgo Trento, Verona
- Mexico (3):
  - CHRISTUS - Latam Hub Excellence and Innovation Center, Monterrey, Nuevo León
  - Centro de Estudios de Investigación Metabólicos y Cardio, Ciudad Madero, Tamaulipas
  - Consultorio de Endocrinología y Pediatría, Puebla City
- Poland (8):
  - Klinika Pediatrii, Endokrynologii, Diabetologii I chorób Metabolicznych, Uniwersyteckiego Szpitala Klinicznego in Wrocław, Wroclaw, Lower Silesian Voivodeship
  - Copernicus Podmiot Leczniczy Sp. z o.o., Gdansk
  - Górnośląskie Centrum Zdrowia Dziecka Im. Św. Jana Pawla II Samodzielny Publiczny Szpital Kliniczny Nr 6 SUM w Katowicach, Katowice
  - UMED Clinical Trials sp. z o.o., Lodz
  - Kliniczny Szpital Wojewodzki nr 2 im. Sw. Jadwigi Krolowej w Rzeszowie, Rzeszów
  - ELIPSA - Elzbieta Lipska praktyka lekarska Osrodek Endokrynologii i Diabetologii Dzieciecej, Stanisławow Pierwszy Nieporet
  - Instytut ''Pomnik - Centrum Zdrowia Dziecka'', Warsaw
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 im. Prof. Szyszko, Zabrze
- Saudi Arabia (5):
  - King Abdulaziz Hospital-Al Ahsa-National Guard, Al Ahsa
  - National Guard Hospital - Jeddah, Jeddah
  - King Khaled University Hospital,King Saud Univ. Med. City, Riyadh
  - King Faisal Specialist Hospital & Research Centre, Riyadh, Riyadh
  - National Guard Hospital_Riyadh, Riyadh
- Sweden (5):
  - Falu Lasarett - Barn- och ungdomsmedicinsk mottagning, Falun
  - Hallands sjukhus Halmstad, Halmstad
  - Barnöverviktsenheten, SUS Malmö, Malmo
  - Sundsvalls sjukhus, Sundsvall
  - Uppsala universitetssjukhus, Uppsala
- United Kingdom (7):
  - Birmingham Children's Hospital, Birmingham
  - University Hospitals Bristol & Weston NHS Foundation Trust, Bristol
  - Leeds Children's Hospital, Leeds
  - Alder Hey Children's Hospital, Liverpool
  - University College Hospital Hospital - Paediatric Services, London
  - Sheffield Children's Hospital, Sheffield
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com